CLINICAL TRIAL: NCT04661150
Title: A Phase II, Randomized Study of Atezolizumab (Anti-PD-L1 Antibody) and Trastuzumab in Combination With Capecitabine and Oxaliplatin (Xelox) in Patients With HER2 Positive Locally Advanced Resectable Gastric Cancer of Adenocarcinoma of Gastroesophageal Junction (GEJ)
Brief Title: A Study of Atezolizumab and Trastuzumab in Combination With Capecitabine and Oxaliplatin in Patients With HER2 Positive Locally Advanced Resectable Gastric Cancer of Adenocarcinoma of Gastroesophageal Junction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML42058
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — atezolizumab; Trastuzumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Atezolizumab plus Trastuzumab with XELOX (Capecitabine + Oxaliplatin) (Experimental): Participants will receive atezolizumab + trastuzumab + XELOX (Capecitabine + Oxaliplatin) for 3 treatment cycles prior to surgery, each cycle is 3 weeks. Following surgery, patrticipants will receive 5 further cycles of this regimen.
  Interventions: Drug: Atezolizumab; Drug: Trastuzumab; Drug: Capecitabine; Drug: Oxaliplatin
- Arm B: Trastuzumab with XELOX (Capecitabine + Oxaliplatin) (Active Comparator): Participants will receive trastuzumab + XELOX (Capecitabine + Oxaliplatin) for 3 treatment cycles prior to surgery, each cycle is 3 weeks. Following surgery, participants will receive 5 further cycles of this regimen.
  Interventions: Drug: Trastuzumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle for 3 cycles prior to surgery and 5 cycles after surgery.
  Other Names: Tecentriq
  Arms: Arm A: Atezolizumab plus Trastuzumab with XELOX (Capecitabine + Oxaliplatin)
Drug: Trastuzumab — Trastuzumab will be administered as an 8 mg/kg IV loading dose and then 6 mg/kg IV on Day 1 of a 21-day cycle for 3 cycles before surgery, and administration will continue after surgery. The first administration of trastuzumab after surgery should also be given at the loading dose of 8 mg/kg.
  Other Names: Herceptin
Drug: Capecitabine — Capecitabine 1000 mg/m^2 will be administered twice orally on Days 1-14, repeated every 3 weeks.
Drug: Oxaliplatin — Oxaliplatin 130 mg/m^2 will be administered by IV on Day 1 of a 21-day cycle.

SUMMARY:
This is a phase II, multicenter, randomized, open-label study designed to evaluate the efficacy and safety of perioperative trastuzumab+XELOX with / without atezolizumab in participants eligible for surgery with locally advanced HER2-positive gastric cancer or adenocarcinoma of GEJ.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric cancer or adenocarcinoma of GEJ
* HER2-positive status defined as either IHC score of 3+ or IHC 2+ with amplification proven by in situ hybridization (ISH) as assessed by local review based on pretreatment endoscopic biopsies.
* Clinical stage at presentation: cT3/T4a/T4b, or N+, M0 as determined by AJCC staging system, 8th edition
* Availability of pretreatment tumor specimen for biomarker analysis by central lab
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy >= 12 weeks
* Adequate hematologic and end-organ function
* For female patients of childbearing potential, agreement (by patient) to remain abstinent (refrain from heterosexual intercourse) or to use highly effective form(s) of contraception during the treatment period and to continue its use for at least i) 5 months after the last dose of atezolizumab, ii) 7 months after the last dose of trastuzumab, or iii) 6 months after the last dose of capecitabine or oxaliplatin, whichever is longer.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Stage IV (metastatic) or unresectable gastric/GEJ cancer determined by investigators
* Prior systemic therapy for treatment of gastric cancer
* History of malignancy other than GC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Cardiopulmonary dysfunction
* Dyspnea at rest
* Active or history of autoimmune disease or immune deficiency with the following exceptions: (a) Patients with a history of autoimmune-mediated hypothyroidism who are on thyroid-replacement hormone are eligible for the study. (b) Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study. (c) Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided allof following conditions are met: (i) Rash must cover < 10% of body surface area (ii) Disease is well controlled at baseline and requires only low-potency topical corticosteroids (iii) No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Active tuberculosis
* Patients with active hepatitis B
* Patients with active hepatitis C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2026-07-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- China (8):
  - Beijing Cancer Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Zhongshan Hospital Fudan University, Shanghai
  - Liaoning Provincial Cancer Hospital, Shengyang
  - First Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Peng Z, Zhang X, Liang H, Zheng Z, Wang Z, Liu H, Hu J, Sun Y, Zhang Y, Yan H, Tong L, Xu J, Ji J, Shen L. Atezolizumab and Trastuzumab Plus Chemotherapy for ERBB2-Positive Locally Advanced Resectable Gastric Cancer: A Randomized Clinical Trial. JAMA Oncol. 2025 Jun 1;11(6):619-624. doi: 10.1001/jamaoncol.2025.0522. PMID 40244574
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin): Participants received atezolizumab + trastuzumab + XELOX (Capecitabine + Oxaliplatin) for 3 treatment cycles prior to surgery, each cycle is 3 weeks. Following surgery, participants received 5 further cycles of this regimen.
- Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin): Participants received trastuzumab + XELOX (Capecitabine + Oxaliplatin) for 3 treatment cycles prior to surgery, each cycle is 3 weeks. Following surgery, participants received 5 further cycles of this regimen.
Period: Overall Study
Arm/Group | Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) | Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin)
Started | 21 | 21
Completed | 0 | 0
Not Completed | 21 | 21
Not completed — Ongoing in study | 19 | 20
Not completed — Refused surgery and for personal reasons. | 0 | 1
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat Population is defined as all participants who were randomly assigned to a treatment, regardless of whether they had surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) | Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin) | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (9.03) | 63.2 (6.28) | 61.5 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Regression (pCR) Rate
Description: pCR is defined as no evidence of vital residual tumor cells on hematoxylin and eosin evaluation of the complete resected gastric/GEJ specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (NAST), which will be reviewed by local pathologist..
Time Frame: Completion of neoadjuvant systemic therapy (up to approximately 16 months)
Population: Intention-to-treat (ITT) population, defined as all participants who were randomly assigned to a treatment, regardless of whether they had surgery.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) | Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin)
Number analyzed (Participants) | 21 | 21
Percentage of Participants | 38.1 [18.1 to 61.6] | 14.3 [3.0 to 36.3]
Statistical Analysis 1: Comparison: Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) vs Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin); Test type: Superiority; p = 0.079, Chi-squared; Treatment difference = 23.8, 90% CI 2-sided [1.3 to 44.7]

2. Secondary Outcome: Event-free Survival (EFS)
Description: Event-free survival (EFS), defined as the time from randomization to the first documented disease recurrence, unequivocal tumor progression determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first.
Time Frame: Randomization to the first documented disease recurrence, unequivocal tumor progression or death from any cause, whichever occurs first (up to approximately 52 months)
Reporting Status: Not Posted, anticipated posting 2027-08

3. Secondary Outcome: Disease-Free Survival (DFS)
Description: Disease-free survival (DFS), defined as the time from surgery to the first documented disease recurrence or death from any cause, whichever occurs first.
Time Frame: Surgery to first documented disease recurrence or death from any cause, whichever occurs first (up to approximately 52 months)
Reporting Status: Not Posted, anticipated posting 2027-08

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS), defined as the time from randomization to death from any cause in all patients.
Time Frame: Randomiation to death from any cause (up to approximately 52 months)
Reporting Status: Not Posted, anticipated posting 2027-08

5. Secondary Outcome: Major Pathologic Response (MPR)
Description: Major pathologic response (MPR), defined as < 10% residual tumor per tumor bed based on evaluation of the resected primary esophagogastric specimen by a local pathologist.
Time Frame: Randomization up to approximately 16 months
Reporting Status: Not Posted, anticipated posting 2027-08

6. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR), defined as the proportion of patients with a complete response (CR) or partial response (PR) during NAST, as determined by the investigator according to RECIST v1.1.
Time Frame: Randomiation to CR or PR during neoadjuvant systemic therapy (up to approximately 16 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) | Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin)
Number analyzed (Participants) | 21 | 21
Percentage of participants | 28.6 [11.3 to 52.2] | 33.3 [14.6 to 57.0]
Statistical Analysis 1: Comparison: Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) vs Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin); Test type: Superiority; p = 0.739, Chi-squared; Treatment difference = -4.8, 90% CI 2-sided [-27.9 to 18.9]

7. Secondary Outcome: R0 Resection Rate
Description: R0 resection rate, defined as the proportion of patients with a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed and/or sampled regional lymph nodes based on evaluation by the local pathologist.
Time Frame: Surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of particpants
Arm/Group | Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) | Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin)
Number analyzed (Participants) | 21 | 21
Percentage of particpants | 95.2 [76.2 to 99.9] | 90.5 [69.6 to 98.8]
Statistical Analysis 1: Comparison: Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) vs Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin); Test type: Superiority; p > 0.999, Fisher Exact; Treatment difference = 4.8, 90% CI 2-sided [-10.9 to 21.4]

8. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Baseline through the end of study (approximately 52 months)
Reporting Status: Not Posted, anticipated posting 2027-08

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 21 March 2022 (up to approximately 12 months)
Description: Serious & other adverse events reported based on safety population, which included patients who received any amount of any component of study treatment. All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized patients.
Arm/Group | Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) | Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin)
All-Cause Mortality (participants affected / at risk) | 2/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 6/21 | 5/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Atezolizumab Plus Trastuzumab With XELOX (Capecitabine + Oxaliplatin) (N=21) | Arm B: Trastuzumab With XELOX (Capecitabine + Oxaliplatin) (N=21)
Nausea (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Platelet count decreased (Investigations) | 4 | 5
Weight decreased (Investigations) | 4 | 1
Bilirubin conjugated increased (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 3 | 3
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood bilirubin unconjugated increased 2 (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 2 | 3
Amylase increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 1
PCO2 decreased (Investigations) | 1 | 0
PO2 decreased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Heart rate decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Asthenia (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 2
Chills (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 2
Peripheral swelling (General disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 2 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 2
Paraesthesia (Nervous system disorders) | 2 | 1
Taste disorder (Nervous system disorders) | 2 | 1
Anaesthesia (Nervous system disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Protein total decreased (Investigations) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT04661150/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT04661150/SAP_001.pdf